CLINICAL TRIAL: NCT05478187
Title: A Wearable Visual Cueing System for Gait Rehabilitation in Parkinson's Disease: a Randomized Controlled Trial.
Brief Title: Wearable Visual Cues in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Habilita, Ospedale di Sarnico (Other)
Responsible Party: Principal Investigator, Michelangelo Bartolo, Director Neurorehabilitation Unit, Habilita S.p.A.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QWalkTrial
Record Dates: First submitted 2022-07-24; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Parkinson Disease; Movement Disorders; Gait Disorders, Neurologic
Keywords: visual cues; sensory cues; gait; balance; rehabilitation; Parkinson's disease; wearable device
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QWalk Study Group (Experimental): 10 individual sessions (5 sessions/week for 2 consecutive weeks). Each session consisted of 60 minutes of conventional physiotherapy plus an additional session of gait training (30 minutes), performed by means of the new wearable cueing system (QWalk)
  Interventions: Device: QWalk Study Group
- Control Group (Active Comparator): 10 individual sessions (5 sessions/week for 2 consecutive weeks). Each session consisted of 60 minutes of conventional physiotherapy plus an additional session of gait training (30 minutes), performed by means of traditional visual cues consisting of stripes on the floor
  Interventions: Other: Traditional visual cues - Control group

INTERVENTIONS:
Device: QWalk Study Group — 10 individual sessions (5 sessions/week for 2 consecutive weeks). Each session consisted of 60 minutes of conventional physiotherapy plus an additional session of gait training (30 minutes), performed by means of the new wearable cueing system (QWalk)
  Other Names: QWalk
  Arms: QWalk Study Group
Other: Traditional visual cues - Control group — 10 individual sessions (5 sessions/week for 2 consecutive weeks). Each session consisted of 60 minutes of conventional physiotherapy plus an additional session of gait training (30 minutes), performed by means of the traditional cues (stripes on the floor)
  Other Names: Traditional cues
  Arms: Control Group

SUMMARY:
One of the most disabling features of Parkinson's disease (PD) is represented by the gait disturbances. Some systematic reviews and meta-analysis have showed that conventional physical therapy might improve gait as well as balance, mobility and functional reach in subjects affected by PD. In addition, several studies and reviews support the effectiveness of external sensory cueing, by means of rhythmic auditory or visual cues, in improving kinematic parameters of gait (gait cadence, stride length, velocity, and postural stability) and the functional performance in people with PD, at least in the short-term. Specifically, cueing refers to the use of temporal or spatial stimuli to regulate movement and facilitate functional performance for individual with motor dysfunction. Basal ganglia act as internal triggers of neuronal activity in the supplementary motor area for well-learned, automatic movement sequences, such as locomotion. This mechanism is damaged in individuals with PD, and external cues may act as an attention resource to compensate the deficient internal rhythm due to basal ganglia dysfunction. Subjects can be coached in concentrating their attention on gait by specific self-prompting instructions or by cues stimulation or a combination of these. Movements generated by the presence of external sensory cues are prompted to use alternative (cortical, parieto-premotor) neuronal pathways which have not been damaged by neuronal degeneration of PD, bypassing the automatic basal ganglia network. Recent studies have provided preliminary evidence that visual cueing based on laser shoes and laser canes may reduce freezing, an established risk for falls, with improvement that can be observed for a variable period of time after rehabilitative intervention. In light of the evidence of effectiveness of cueing, developing wearable devices able to generate cues that match with step and that are effective, easy to use and low cost, would be challenging but very appropriate. The aim of this study was to investigate the non-inferiority of a wearable device producing visual cues (Q-Walk system, QUICKLYPRO s.r.l., Bergamo, Italy) in order to improve gait and balance PD patients, compared to a conventional training (stripes on the floor).

DETAILED DESCRIPTION:
All patients consecutively referred to the Neurorehabilitation Unit of HABILITA between 1st November 2019 and 31th December 2021 were screened. Patient were admitted for outpatients rehabilitation. All particpants could walk independently without walking device. All patients were taking oral administration of levodopa, dopamine agonists, or both, and were evaluated in ON phase.

All the patients gave their written informed consent to take part in the study. The study was approved by the Local Ethics Committee of Bergamo (Reg. Sper. n. 178/19, 11/10/2019) and was carried out in accordance with The Code of Ethics of the World Medical Association (Declaration of Helsinki) for experiments involving humans.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic PD (defined by the UK Brain Bank Criteria);
* absence of cognitive impairment (Mini-Mental State Examination score ≥ 24);
* Hoehn & Yahr stage II-IV; mild to severe gait disturbance with score ≥2 at the Unified Parkinson's Disease Rating Scale (UPDRS) motor section III;
* stable drug usage since at least 3 weeks.

Exclusion Criteria:

* past history or current presence of neurological conditions other than PD;
* orthopedic or visual disturbances severely impairing walking ability;
* previous deep brain stimulation or other neurosurgery;
* participation in a rehabilitation program within 2 months before the trial and previous use of cues for gait rehabilitation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
mean gait speed (m/s) change | Change from baseline (Time 0) at the end of the intervention (2 weeks - Time 1) and at the followup (3 months - Time 2)
  Distance covered by the body in the unit of time
step length (m) change | Change from baseline (Time 0) at the end of the intervention (2 weeks - Time 1) and at the followup (3 months - Time 2)
  Distance measured from the heel print of one foot to the heel print of the other foot
cadence (step/min) change | Change from baseline (Time 0) at the end of the intervention (2 weeks - Time 1) and at the followup (3 months - Time 2)
  time of steps per unit time
stance phase duration (%) change | Change from baseline (Time 0) at the end of the intervention (2 weeks - Time 1) and at the followup (3 months - Time 2)
  time interval between two consecutive foot strikes of the same lower limb expressed as a percentage of the stride duration
double support phase duration (%) change | Change from baseline (Time 0) at the end of the intervention (2 weeks - Time 1) and at the followup (3 months - Time 2)
  Time of the sub-phase between heel contact of the phase to contralateral foot-off

SECONDARY OUTCOMES:
CoP sway length (statokinesigram) (mm) change | Change from baseline (Time 0) at the end of the intervention (2 weeks - Time 1) and at the followup (3 months - Time 2)
  The projection onto a 2-dimensional space of the trajectory of the centre of pressure (COP) of a person during erect stance
mean CoP position along the anteroposterior direction (Eyes Open) change | Change from baseline (Time 0) at the end of the intervention (2 weeks - Time 1) and at the followup (3 months - Time 2)
  the centroid of all the external forces acting on the plantar surface of the foot
mean CoP position along the mediolateral direction (Eyes Open) change | Change from baseline (Time 0) at the end of the intervention (2 weeks - Time 1) and at the followup (3 months - Time 2)
  the centroid of all the external forces acting on the plantar surface of the foot
mean CoP position along the anteroposterior direction (Eyes Closed) change | Change from baseline (Time 0) at the end of the intervention (2 weeks - Time 1) and at the followup (3 months - Time 2)
  the centroid of all the external forces acting on the plantar surface of the foot
mean CoP position along the mediolateral direction (Eyes Closed) change | Change from baseline (Time 0) at the end of the intervention (2 weeks - Time 1) and at the followup (3 months - Time 2)
  the centroid of all the external forces acting on the plantar surface of the foot

CONTACTS AND LOCATIONS:
Overall Officials: Michelangelo Bartolo, Md, PhD, Principal Investigator — Habilita Zingonia
Locations (1):
- Habilita Zingonia, Ciserano, Bergamo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boonstra TA, van der Kooij H, Munneke M, Bloem BR. Gait disorders and balance disturbances in Parkinson's disease: clinical update and pathophysiology. Curr Opin Neurol. 2008 Aug;21(4):461-71. doi: 10.1097/WCO.0b013e328305bdaf. PMID 18607208
- [Background] Moustafa AA, Chakravarthy S, Phillips JR, Crouse JJ, Gupta A, Frank MJ, Hall JM, Jahanshahi M. Interrelations between cognitive dysfunction and motor symptoms of Parkinson's disease: behavioral and neural studies. Rev Neurosci. 2016 Jul 1;27(5):535-48. doi: 10.1515/revneuro-2015-0070. PMID 26982614
- [Background] Cassimatis C, Liu KP, Fahey P, Bissett M. The effectiveness of external sensory cues in improving functional performance in individuals with Parkinson's disease: a systematic review with meta-analysis. Int J Rehabil Res. 2016 Sep;39(3):211-8. doi: 10.1097/MRR.0000000000000171. PMID 27119224
- [Background] De Nunzio A, Zucchella C, Spicciato F, Tortola P, Vecchione C, Pierelli F, Bartolo M. Biofeedback rehabilitation of posture and weightbearing distribution in stroke: a center of foot pressure analysis. Funct Neurol. 2014 Apr-Jun;29(2):127-34. PMID 25306123
- [Background] Nonnekes J, Nieuwboer A. Towards Personalized Rehabilitation for Gait Impairments in Parkinson's Disease. J Parkinsons Dis. 2018;8(s1):S101-S106. doi: 10.3233/JPD-181464. PMID 30584154